CLINICAL TRIAL: NCT00798876
Title: Comparison Study of a Low-Fat Diet Supplemented With Fish Oil and a Standard Western Diet in Individuals With Prostate Cancer
Brief Title: Low-Fat Fish Oil Diet for Prostate Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-07-026; P50CA092131-01A1 (NIH); 11-002610 (Other: JCCC); NCT00836615 (obsolete NCT alias)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fish Oils; Diet, Western; Diet, Fat-Restricted; Independent Medical Evaluation; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Western Diet (Placebo Comparator): Subjects will be asked to consume a standard Western Diet for 4 weeks. For the 4-week period, subjects will be provided with all food and beverages. Subjects will also undergo a medical examination, dietary interview, blood draw, and radical prostatectomy(as part of standard of care).
  Interventions: Dietary Supplement: Western Diet; Other: Medical Examination; Other: Dietary Interview; Other: Blood Draw; Procedure: Radical Prostatectomy
- Low-Fat Diet (Experimental): Subjects will be asked to consume a low fat diet with fish oil and vitamin E supplements for 4 weeks. For the 4-week period, subjects will be provided with all food and beverages. Subjects will also undergo a medical examination, dietary interview, blood draw, and radical prostatectomy(as part of standard of care).
  Interventions: Dietary Supplement: Fish Oil; Dietary Supplement: Vitamin E supplement; Dietary Supplement: Low-Fat Diet; Other: Medical Examination; Other: Dietary Interview; Other: Blood Draw; Procedure: Radical Prostatectomy

INTERVENTIONS:
Dietary Supplement: Fish Oil — Subjects will be asked to take 10 grams of fish oil per day for 4 weeks.
  Arms: Low-Fat Diet
Dietary Supplement: Vitamin E supplement — Subjects will be asked to take 800 International Units per day of Vitamin E for 4 weeks.
  Arms: Low-Fat Diet
Dietary Supplement: Western Diet — Subjects will be provided with a standard western diet, food and beverages, to consume during their 4 week participation in this study.
  Arms: Standard Western Diet
Dietary Supplement: Low-Fat Diet — Subjects will be provided with a low-fat diet (food and beverages) for their 4 week participation in this study.
  Arms: Low-Fat Diet
Other: Medical Examination — Subjects will have a routine medical exam.
Other: Dietary Interview — Subjects will meet with the study nutritionist and have their current diet evaluated. Subjects will also undergo a test (bioimpedance) to estimate their body fat, lean weight, and the rate at which their body burns fat.
Other: Blood Draw — 40 mL of blood will be drawn from subjects to measure PSA, fatty acids, insulin and various hormones.
Procedure: Radical Prostatectomy — Subjects will undergo a radical prostatectomy as part of their standard of care.

SUMMARY:
Studies on patterns of how many men get prostate cancer in other countries show that environment contributes to the high incidence of prostate cancer in the United States. Epidemiology studies suggest that this influence may be reduced by the diet of men at risk of getting prostate cancer. Although the exact nature of the effects of diet are not completely known, the amount of fat eaten appears to affect the number of men who get prostate cancer. The type of fat also seems to matter. Eating more of a type of fat called omega-3 polyunsaturated fat is associated with decreased prostate cancer risk. Omega-3 fat comes from fish and is quite different from the type of fat from animals and vegetables (omega-6 fat). Because the exact mechanism of this reduction in prostate cancer risk is not known, no blood test indications, called markers, have been discovered that would show the effect working.

Study doctors designed this study to try to find markers in the blood tests of men who have prostate cancer, and to find out if a diet supplemented with omega-3 type fat from fish oil helps reduce those markers, hence indicating that it helps reduce the cancer in these men. These men will be compared to men with prostate cancer whose diets do not contain the fish-oil fat.

The men chosen will have prostate cancer and be scheduled for operations to have their prostate glands removed. They will be chosen randomly to be given the fish-oil diet or a regular Western diet for comparison for 4 to 8 weeks. Their blood will be checked at the beginning of the diet. After the 4-to-8-week period, they will have their operations. Their blood will be checked again and a sample of their removed prostate will be examined to tell if the diet had any effect on the cancer and its markers.

DETAILED DESCRIPTION:
1. To establish and validate intermediate biomarkers for prostate cancer prevention trials by conducting a dietary intervention trial of a low-fat diet with omega-3 fatty acid supplements in men undergoing radical prostatectomy. In initial trials it was feasible to intervene with diet and obtain tissue and serum for bioassay and biomarker development. This aim is to study the effect a low-fat, high omega-3 diet has on serum and tissue biomarkers from patients who have prostatectomies for prostate cancer. Ultimately, we hope to identify and validate intermediate markers of efficacy for large-scale dietary prevention trials.
2. To establish and validate insulin growth factor-1 (IGF-1) and insulin growth factor binding proteins (IGFBP) as relevant intermediate biomarkers for prostate cancer prevention trials. IGF-1 is a peptide growth factor that is important to the growth and progression of prostate cancer. To our knowledge, no prospective dietary intervention studies have evaluated the effect of a low-fat diet with omega-3 fatty acid supplements on IGF-1 and IGFBPs, and their potential to serve as relevant intermediate markers for low-fat dietary intervention trials for prostate cancer prevention.
3. To establish and validate serum and tissue fatty acids as relevant intermediate biomarkers for prostate cancer prevention trials. We will evaluate if men randomized to a low-fat, fish-oil-supplemented diet have increased serum ratios of omega-3:omega-6 fatty acids compared with men randomized to a control Western diet before radical prostatectomy. We also will study if patients in the low-fat, fish oil arm have increased ratios of membrane omega-3:omega-6 fatty acids as well as decreased COX-2 and decreased PGE-2 levels in benign and malignant tissue and in visceral fat. If so, it will proved further evidence to support the potential of low-fat fish oil diets for prostate cancer prevention. If serum omega-3:omega-6 ratios correlate with changes in COX-2 and PGE-2 in tissues, then serum omea-3:omega-6 ratios may be useful for monitoring activity and efficacy of low-fat fish-oil-supplemented diets in future trials.

ELIGIBILITY:
Eligibility Criteria:

* Patient consents to participate.
* Medically able to receive and comply with the diet.
* Lives near enough for counseling and follow-up.
* Has elected to have operation to remove prostate.
* Agrees to stop diet or vitamin supplements or herbal supplements for 1 week before the study begins.
* Patient able to stop taking aspirin, COX-2 inhibitors, and other anti-inflammatory medications for 1 week before study start.
* Patient able to safely stop taking fish oil capsules 2 weeks before the diet starts.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2001-12-18 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
check for insulin growth factor-1 (IGF-1) and insulin growth factor binding proteins (IGFBP) as relevant intermediate biomarkers for prostate cancer | 4 weeks

SECONDARY OUTCOMES:
Check serum and tissue fatty acids as relevant intermediate biomarkers for prostate cancer | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Aronson, MD, Principal Investigator — UCLA and Western Los Angles VA
Locations (2):
- United States (2):
  - West Los Angeles VA, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California

REFERENCES:
- [Background] Landis SH, Murray T, Bolden S, Wingo PA. Cancer statistics, 1999. CA Cancer J Clin. 1999 Jan-Feb;49(1):8-31, 1. doi: 10.3322/canjclin.49.1.8. PMID 10200775
- [Background] Parkin DM, Pisani P, Ferlay J. Global cancer statistics. CA Cancer J Clin. 1999 Jan-Feb;49(1):33-64, 1. doi: 10.3322/canjclin.49.1.33. PMID 10200776
- [Background] Muir CS, Nectoux J, Staszewski J. The epidemiology of prostatic cancer. Geographical distribution and time-trends. Acta Oncol. 1991;30(2):133-40. doi: 10.3109/02841869109092336. PMID 2029395
- [Background] Yatani R, Kusano I, Shiraishi T, Hayashi T, Stemmermann GN. Latent prostatic carcinoma: pathological and epidemiological aspects. Jpn J Clin Oncol. 1989 Dec;19(4):319-26. PMID 2691730
- [Background] Shimizu H, Ross RK, Bernstein L, Yatani R, Henderson BE, Mack TM. Cancers of the prostate and breast among Japanese and white immigrants in Los Angeles County. Br J Cancer. 1991 Jun;63(6):963-6. doi: 10.1038/bjc.1991.210. PMID 2069852
- [Background] Stellman SD, Wang QS. Cancer mortality in Chinese immigrants to New York City. Comparison with Chinese in Tianjin and with United States-born whites. Cancer. 1994 Feb 15;73(4):1270-5. doi: 10.1002/1097-0142(19940215)73:43.0.co;2-y. PMID 8313330
- [Background] Cook LS, Goldoft M, Schwartz SM, Weiss NS. Incidence of adenocarcinoma of the prostate in Asian immigrants to the United States and their descendants. J Urol. 1999 Jan;161(1):152-5. PMID 10037388
- [Background] Whittemore AS, Kolonel LN, Wu AH, John EM, Gallagher RP, Howe GR, Burch JD, Hankin J, Dreon DM, West DW, et al. Prostate cancer in relation to diet, physical activity, and body size in blacks, whites, and Asians in the United States and Canada. J Natl Cancer Inst. 1995 May 3;87(9):652-61. doi: 10.1093/jnci/87.9.652. PMID 7752270
- [Background] Boyle P, Levi F, Lucchini F, La Vecchia C, Kevi R [corrected to Levi F], Lucchuni F [corrected to Lucchini F]. Trends in diet-related cancers in Japan: a conundrum? Lancet. 1993 Sep 18;342(8873):752. doi: 10.1016/0140-6736(93)91748-b. No abstract available. PMID 8103867
- [Background] Wynder EL, Fujita Y, Harris RE, Hirayama T, Hiyama T. Comparative epidemiology of cancer between the United States and Japan. A second look. Cancer. 1991 Feb 1;67(3):746-63. doi: 10.1002/1097-0142(19910201)67:33.0.co;2-1. PMID 1985768
- [Background] Giovannucci E, Rimm EB, Colditz GA, Stampfer MJ, Ascherio A, Chute CG, Willett WC. A prospective study of dietary fat and risk of prostate cancer. J Natl Cancer Inst. 1993 Oct 6;85(19):1571-9. doi: 10.1093/jnci/85.19.1571. PMID 8105097
- [Background] West DW, Slattery ML, Robison LM, French TK, Mahoney AW. Adult dietary intake and prostate cancer risk in Utah: a case-control study with special emphasis on aggressive tumors. Cancer Causes Control. 1991 Mar;2(2):85-94. doi: 10.1007/BF00053126. PMID 1873441
- [Background] Kolonel LN, Yoshizawa CN, Hankin JH. Diet and prostatic cancer: a case-control study in Hawaii. Am J Epidemiol. 1988 May;127(5):999-1012. doi: 10.1093/oxfordjournals.aje.a114903. PMID 3358418
- [Background] Fradet Y, Meyer F, Bairati I, Shadmani R, Moore L. Dietary fat and prostate cancer progression and survival. Eur Urol. 1999;35(5-6):388-91. doi: 10.1159/000019913. PMID 10325493
- [Background] Wang Y, Corr JG, Thaler HT, Tao Y, Fair WR, Heston WD. Decreased growth of established human prostate LNCaP tumors in nude mice fed a low-fat diet. J Natl Cancer Inst. 1995 Oct 4;87(19):1456-62. doi: 10.1093/jnci/87.19.1456. PMID 7545759
- [Background] Severson RK, Nomura AM, Grove JS, Stemmermann GN. A prospective study of demographics, diet, and prostate cancer among men of Japanese ancestry in Hawaii. Cancer Res. 1989 Apr 1;49(7):1857-60. PMID 2924323
- [Background] Hsing AW, McLaughlin JK, Schuman LM, Bjelke E, Gridley G, Wacholder S, Chien HT, Blot WJ. Diet, tobacco use, and fatal prostate cancer: results from the Lutheran Brotherhood Cohort Study. Cancer Res. 1990 Nov 1;50(21):6836-40. PMID 2208150
- [Background] Kris-Etherton PM, Taylor DS, Yu-Poth S, Huth P, Moriarty K, Fishell V, Hargrove RL, Zhao G, Etherton TD. Polyunsaturated fatty acids in the food chain in the United States. Am J Clin Nutr. 2000 Jan;71(1 Suppl):179S-88S. doi: 10.1093/ajcn/71.1.179S. PMID 10617969
- [Background] Baghurst KI, Crawford DA, Worsley A, Record SJ. The Victorian Nutrition Survey--intakes and sources of dietary fats and cholesterol in the Victorian population. Med J Aust. 1988 Jul 4;149(1):12-5, 18-20. doi: 10.5694/j.1326-5377.1988.tb120476.x. PMID 3386562
- [Background] Sugano M, Hirahara F. Polyunsaturated fatty acids in the food chain in Japan. Am J Clin Nutr. 2000 Jan;71(1 Suppl):189S-96S. doi: 10.1093/ajcn/71.1.189S. PMID 10617970
- [Background] Mishina T, Watanabe H, Araki H, Nakao M. Epidemiological study of prostatic cancer by matched-pair analysis. Prostate. 1985;6(4):423-36. doi: 10.1002/pros.2990060411. PMID 4088954
- [Background] Godley PA, Campbell MK, Gallagher P, Martinson FE, Mohler JL, Sandler RS. Biomarkers of essential fatty acid consumption and risk of prostatic carcinoma. Cancer Epidemiol Biomarkers Prev. 1996 Nov;5(11):889-95. PMID 8922296
- [Background] Kobayashi M, Sasaki S, Hamada GS, Tsugane S. Serum n-3 fatty acids, fish consumption and cancer mortality in six Japanese populations in Japan and Brazil. Jpn J Cancer Res. 1999 Sep;90(9):914-21. doi: 10.1111/j.1349-7006.1999.tb00835.x. PMID 10551318
- [Background] Norrish AE, Skeaff CM, Arribas GL, Sharpe SJ, Jackson RT. Prostate cancer risk and consumption of fish oils: a dietary biomarker-based case-control study. Br J Cancer. 1999 Dec;81(7):1238-42. doi: 10.1038/sj.bjc.6690835. PMID 10584888
- [Background] Schuurman AG, van den Brandt PA, Dorant E, Brants HA, Goldbohm RA. Association of energy and fat intake with prostate carcinoma risk: results from The Netherlands Cohort Study. Cancer. 1999 Sep 15;86(6):1019-27. PMID 10491529
- [Background] Zhou JR, Blackburn GL. Bridging animal and human studies: what are the missing segments in dietary fat and prostate cancer? Am J Clin Nutr. 1997 Dec;66(6 Suppl):1572S-1580S. doi: 10.1093/ajcn/66.6.1572S. PMID 9394717
- [Background] Rose DP, Connolly JM. Effects of fatty acids and eicosanoid synthesis inhibitors on the growth of two human prostate cancer cell lines. Prostate. 1991;18(3):243-54. doi: 10.1002/pros.2990180306. PMID 2020620
- [Background] Pandalai PK, Pilat MJ, Yamazaki K, Naik H, Pienta KJ. The effects of omega-3 and omega-6 fatty acids on in vitro prostate cancer growth. Anticancer Res. 1996 Mar-Apr;16(2):815-20. PMID 8687134
- [Background] Rose DP, Cohen LA. Effects of dietary menhaden oil and retinyl acetate on the growth of DU 145 human prostatic adenocarcinoma cells transplanted into athymic nude mice. Carcinogenesis. 1988 Apr;9(4):603-5. doi: 10.1093/carcin/9.4.603. PMID 3356068
- [Background] Iwamura M, Sluss PM, Casamento JB, Cockett AT. Insulin-like growth factor I: action and receptor characterization in human prostate cancer cell lines. Prostate. 1993;22(3):243-52. doi: 10.1002/pros.2990220307. PMID 8488157
- [Background] Yu H, Rohan T. Role of the insulin-like growth factor family in cancer development and progression. J Natl Cancer Inst. 2000 Sep 20;92(18):1472-89. doi: 10.1093/jnci/92.18.1472. PMID 10995803
- [Background] Chan JM, Stampfer MJ, Giovannucci E, Gann PH, Ma J, Wilkinson P, Hennekens CH, Pollak M. Plasma insulin-like growth factor-I and prostate cancer risk: a prospective study. Science. 1998 Jan 23;279(5350):563-6. doi: 10.1126/science.279.5350.563. PMID 9438850
- [Background] Wolk A, Mantzoros CS, Andersson SO, Bergstrom R, Signorello LB, Lagiou P, Adami HO, Trichopoulos D. Insulin-like growth factor 1 and prostate cancer risk: a population-based, case-control study. J Natl Cancer Inst. 1998 Jun 17;90(12):911-5. doi: 10.1093/jnci/90.12.911. PMID 9637140
- [Background] Mantzoros CS, Tzonou A, Signorello LB, Stampfer M, Trichopoulos D, Adami HO. Insulin-like growth factor 1 in relation to prostate cancer and benign prostatic hyperplasia. Br J Cancer. 1997;76(9):1115-8. doi: 10.1038/bjc.1997.520. PMID 9365156
- [Background] Kaplan PJ, Mohan S, Cohen P, Foster BA, Greenberg NM. The insulin-like growth factor axis and prostate cancer: lessons from the transgenic adenocarcinoma of mouse prostate (TRAMP) model. Cancer Res. 1999 May 1;59(9):2203-9. PMID 10232609
- [Background] Mukherjee P, Sotnikov AV, Mangian HJ, Zhou JR, Visek WJ, Clinton SK. Energy intake and prostate tumor growth, angiogenesis, and vascular endothelial growth factor expression. J Natl Cancer Inst. 1999 Mar 17;91(6):512-23. doi: 10.1093/jnci/91.6.512. PMID 10088621
- [Background] Dunn SE, Kari FW, French J, Leininger JR, Travlos G, Wilson R, Barrett JC. Dietary restriction reduces insulin-like growth factor I levels, which modulates apoptosis, cell proliferation, and tumor progression in p53-deficient mice. Cancer Res. 1997 Nov 1;57(21):4667-72. PMID 9354418
- [Background] Ferry RJ Jr, Katz LE, Grimberg A, Cohen P, Weinzimer SA. Cellular actions of insulin-like growth factor binding proteins. Horm Metab Res. 1999 Feb-Mar;31(2-3):192-202. doi: 10.1055/s-2007-978719. PMID 10226802
- [Background] Thissen JP, Ketelslegers JM, Underwood LE. Nutritional regulation of the insulin-like growth factors. Endocr Rev. 1994 Feb;15(1):80-101. doi: 10.1210/edrv-15-1-80. PMID 8156941
- [Background] Donaghy AJ, Baxter RC. Insulin-like growth factor bioactivity and its modification in growth hormone resistant states. Baillieres Clin Endocrinol Metab. 1996 Jul;10(3):421-46. doi: 10.1016/s0950-351x(96)80560-x. PMID 8853449
- [Background] Nam SY, Lee EJ, Kim KR, Cha BS, Song YD, Lim SK, Lee HC, Huh KB. Effect of obesity on total and free insulin-like growth factor (IGF)-1, and their relationship to IGF-binding protein (BP)-1, IGFBP-2, IGFBP-3, insulin, and growth hormone. Int J Obes Relat Metab Disord. 1997 May;21(5):355-9. doi: 10.1038/sj.ijo.0800412. PMID 9152736
- [Background] Nyomba BL, Berard L, Murphy LJ. Free insulin-like growth factor I (IGF-I) in healthy subjects: relationship with IGF-binding proteins and insulin sensitivity. J Clin Endocrinol Metab. 1997 Jul;82(7):2177-81. doi: 10.1210/jcem.82.7.4070. PMID 9215291
- [Background] Scacchi M, Pincelli AI, Cavagnini F. Growth hormone in obesity. Int J Obes Relat Metab Disord. 1999 Mar;23(3):260-71. doi: 10.1038/sj.ijo.0800807. PMID 10193871
- [Background] Grimberg A, Cohen P. Role of insulin-like growth factors and their binding proteins in growth control and carcinogenesis. J Cell Physiol. 2000 Apr;183(1):1-9. doi: 10.1002/(SICI)1097-4652(200004)183:13.0.CO;2-J. PMID 10699960
- [Background] Signorello LB, Brismar K, Bergstrom R, Andersson SO, Wolk A, Trichopoulos D, Adami HO. Insulin-like growth factor-binding protein-1 and prostate cancer. J Natl Cancer Inst. 1999 Nov 17;91(22):1965-7. doi: 10.1093/jnci/91.22.1965. No abstract available. PMID 10564682
- [Background] Bagga D, Capone S, Wang HJ, Heber D, Lill M, Chap L, Glaspy JA. Dietary modulation of omega-3/omega-6 polyunsaturated fatty acid ratios in patients with breast cancer. J Natl Cancer Inst. 1997 Aug 6;89(15):1123-31. doi: 10.1093/jnci/89.15.1123. PMID 9262250
- [Background] Hansen HS. Dietary essential fatty acids and in vivo prostaglandin production in mammals. World Rev Nutr Diet. 1983;42:102-34. doi: 10.1159/000408352. No abstract available. PMID 6375159
- [Background] Karmali RA. Eicosanoids in neoplasia. Prev Med. 1987 Jul;16(4):493-502. doi: 10.1016/0091-7435(87)90063-6. PMID 3114735
- [Background] Culp BR, Titus BG, Lands WE. Inhibition of prostaglandin biosynthesis by eicosapentaenoic acid. Prostaglandins Med. 1979 Nov;3(5):269-78. doi: 10.1016/0161-4630(79)90068-5. PMID 121610
- [Background] Rose DP, Connolly JM. Dietary fat, fatty acids and prostate cancer. Lipids. 1992 Oct;27(10):798-803. doi: 10.1007/BF02535853. PMID 1435098
- [Background] Levy GN. Prostaglandin H synthases, nonsteroidal anti-inflammatory drugs, and colon cancer. FASEB J. 1997 Mar;11(4):234-47. PMID 9068612
- [Background] Marnett LJ. Prostaglandin synthase-mediated metabolism of carcinogens and a potential role for peroxyl radicals as reactive intermediates. Environ Health Perspect. 1990 Aug;88:5-12. doi: 10.1289/ehp.90885. PMID 2125560
- [Background] Ablin RJ, Shaw MW. Prostaglandin modulation of prostate tumor growth and metastases. Anticancer Res. 1986 Mar-Apr;6(2):327-8. No abstract available. PMID 3486627
- [Background] Smith BJ, Wills MR, Savory J. Prostaglandins and cancer. Ann Clin Lab Sci. 1983 Sep-Oct;13(5):359-65. PMID 6357045
- [Background] Rubenstein M, Shaw MW, McKiel CF, Ray PS, Guinan PD. Immunoregulatory markers in rats carrying Dunning R3327 H, G, or MAT-LyLu prostatic adenocarcinoma variants. Cancer Res. 1987 Jan 1;47(1):178-82. PMID 3491674
- [Background] Shaw MW, Ablin RJ, Ray P, Rubenstein M, Guinan PD, McKiel CF. Immunobiology of the Dunning R-3327 rat prostate adenocarcinoma sublines: plasma and tumor effusion prostaglandins. Am J Reprod Immunol Microbiol. 1985 Jul;8(3):77-9. doi: 10.1111/j.1600-0897.1985.tb00312.x. PMID 3861106
- [Background] Vane JR, Bakhle YS, Botting RM. Cyclooxygenases 1 and 2. Annu Rev Pharmacol Toxicol. 1998;38:97-120. doi: 10.1146/annurev.pharmtox.38.1.97. PMID 9597150
- [Background] Tjandrawinata RR, Dahiya R, Hughes-Fulford M. Induction of cyclo-oxygenase-2 mRNA by prostaglandin E2 in human prostatic carcinoma cells. Br J Cancer. 1997;75(8):1111-8. doi: 10.1038/bjc.1997.192. PMID 9099957
- [Background] Gupta S, Srivastava M, Ahmad N, Bostwick DG, Mukhtar H. Over-expression of cyclooxygenase-2 in human prostate adenocarcinoma. Prostate. 2000 Jan;42(1):73-8. doi: 10.1002/(sici)1097-0045(20000101)42:13.0.co;2-g. PMID 10579801
- [Background] Hwang D, Scollard D, Byrne J, Levine E. Expression of cyclooxygenase-1 and cyclooxygenase-2 in human breast cancer. J Natl Cancer Inst. 1998 Mar 18;90(6):455-60. doi: 10.1093/jnci/90.6.455. PMID 9521170
- [Background] Tsujii M, Kawano S, DuBois RN. Cyclooxygenase-2 expression in human colon cancer cells increases metastatic potential. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):3336-40. doi: 10.1073/pnas.94.7.3336. PMID 9096394
- [Background] Kirschenbaum A, Klausner AP, Lee R, Unger P, Yao S, Liu XH, Levine AC. Expression of cyclooxygenase-1 and cyclooxygenase-2 in the human prostate. Urology. 2000 Oct 1;56(4):671-6. doi: 10.1016/s0090-4295(00)00674-9. PMID 11018637
- [Background] Yoshimura R, Sano H, Masuda C, Kawamura M, Tsubouchi Y, Chargui J, Yoshimura N, Hla T, Wada S. Expression of cyclooxygenase-2 in prostate carcinoma. Cancer. 2000 Aug 1;89(3):589-96. PMID 10931458
- [Background] Norrish AE, Jackson RT, McRae CU. Non-steroidal anti-inflammatory drugs and prostate cancer progression. Int J Cancer. 1998 Aug 12;77(4):511-5. doi: 10.1002/(sici)1097-0215(19980812)77:43.0.co;2-x. PMID 9679750
- [Background] Bucher C, Jordan P, Nickeleit V, Torhorst J, Mihatsch MJ. Relative risk of malignant tumors in analgesic abusers. Effects of long-term intake of aspirin. Clin Nephrol. 1999 Feb;51(2):67-72. PMID 10069640
- [Background] Magoha GA. Ten years experience with chronic prostatitis in Africans. East Afr Med J. 1996 Mar;73(3):176-8. PMID 8698016
- [Background] Lepage G, Roy CC. Direct transesterification of all classes of lipids in a one-step reaction. J Lipid Res. 1986 Jan;27(1):114-20. PMID 3958609
- [Background] Shin BC, Ebner KE, Hudson BG, Carraway KL. Membrane glycoprotein differences between normal lactating mammary tissue and the R3230 AC mammary tumor. Cancer Res. 1975 May;35(5):1135-40. PMID 123479
- [Background] Feldman JM, Hilf R. A role of estrogens and insulin binding in the dietary lipid alteration of R3230AC mammary carcinoma growth in rats. Cancer Res. 1985 May;45(5):1964-72. PMID 3886127
- [Background] Schuman LM, Mandel JS, Radke A, et al: Some elected features of the epidemiology of prostatic cancer: Minneapolis-St. Paul, Minnesota case-control study, 1976-1979. In: Magnus K, ed. Trends in cancer incidence. Washington DC: Hemisphere, 345-354, 1982.